CLINICAL TRIAL: NCT04994938
Title: The Development and Implementation of a Peer-Led Diet and Exercise Intervention in Older Urban Dwelling Veterans With Dysmobility
Brief Title: Peer-Led Diet and Exercise Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E3739-P; RX003739-01A1 (Other Grant/Funding Number: Veteran Affairs Rehabilitation R&D Service)
Record Dates: First submitted 2021-07-27; First posted 2021-08-06 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Physical Activity; Peer Leaders; Diet Quality
Keywords: Diet Quality; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peer led diet and exercise intervention (Experimental): participation in two-times per week diet and exercise peer led interventions.
  Interventions: Other: Diet Intervention; Other: Exercise Intervention

INTERVENTIONS:
Other: Diet Intervention — Participants will engage in discussions about healthy eating one time per week led by a trained peer leader for 12-weeks.
Other: Exercise Intervention — Participants will participate in a group exercise session led by a trained peer leader 2-times per week for 12-weeks.

SUMMARY:
The majority of older Veterans do not meet the minimum healthy diet or physical activity recommendations, despite known benefits. Identifying novel ways to increase adherence to rehabilitation programs that improve dietary quality and physical activity may reduce the risk of disability in older Veterans. Peer-based interventions may be one method to facilitate lasting behavioral change since peers often share a common culture and knowledge about the problems that their community experiences. The investigators propose to develop and evaluate a novel peer-led diet and exercise intervention that targets older Veterans with multiple chronic health conditions. Successful development and pilot of this intervention will provide the preliminary data for a larger multisite trial focused on the use of peer-led interventions to improve long-term compliance to lifestyle interventions in older Veterans.

DETAILED DESCRIPTION:
Over the next ten years the share of Veterans age 65+ years will increase to over 50% of the total Veteran population. The ability to safely maintain mobility with aging is critical. Older Veterans with multiple chronic health conditions are more likely to experience mobility decline and report reduced physical activity levels and poor dietary quality. While a multitude of interventions have attempted to address poor diet and physical inactivity in older adults; most have utilized resource-intensive professionally led diet OR exercise interventions, and few have focused on the unique needs of older Veterans. Peer support offers a potentially low-cost, easily scalable approach to encourage long-term dietary and physical activity change.

In this proposal the investigators seek to develop and pilot a 12-week peer-led lifestyle intervention that targets older Veterans with multiple chronic health conditions and dysmobility, in two diverse urban areas with a high percentage of underrepresented minority Veteran populations (Baltimore, MD and San Antonio, TX). The investigators will develop a theory-driven, peer-led nutrition and exercise intervention tailored for older Veterans with dysmobility. The investigators will also determine the feasibility and acceptability of the peer-led intervention as well as the estimated magnitude and potential impact on selected outcomes (i.e diet quality and mobility) in older Veterans with dysmobility and multiple chronic health conditions.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported difficulty in at least one of the following activities: Walking quickly across the street, walking one mile, ascending one flight of stairs, rising from a chair without using arms
* Self-reports at least two chronic medical conditions such as hypertension, diabetes, hyperlipidemia, or coronary artery disease
* Speaks English

Exclusion Criteria:

* high cardiovascular risk
* using home oxygen
* contraindications to an exercise intervention
* dementia
* regular exercise participation
* current participation in a weight loss intervention
* acute psychosis, major depression, or behavior that preventions group interaction

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Endurance | 12-weeks
  Cardiovascular endurance will be assessed with the distance covered during a six-minute walk test. The distance covered from baseline will be compared to post 12-week intervention.
Diet Quality | 12-weeks
  Food records will be gathered and analyzed using the automated self-administered recall system (ASA24) to evaluate diet quality. Results from baseline will be compared to those after 12 weeks of intervention.

SECONDARY OUTCOMES:
Mobility | 12-weeks
  The number of time and individuals can rise from a chair-without using their arms during a 30-second time period will be recorded and used as a measure of mobility. Results from baseline will be compared to those after 12-weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Odessa R. Addison, PhD DPT, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (2):
- United States (2):
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robbins RN, Serra MC, Kilpela LS, Parker EA, Jiwani R, Addison O. Intervention in Older Urban-Dwelling Veterans With Dysmobility: Protocol for a Pilot Feasibility Clinical Trial. JMIR Res Protoc. 2022 Jul 13;11(7):e39192. doi: 10.2196/39192. PMID 35830251

DOCUMENTS (1):
  • Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT04994938/ICF_000.pdf